Stop-NSBB ICF English V1.2 16May2024

Stop-NSBB Study Patient Information Sheet and Informed Consent Form (Version 1.2)

Study title: Assessing the safety of discontinuing non-selective beta-blockers in cirrhotic patients

with managed primary aetiological factors according to Baveno VII consensus

**Principal investigator:** Dr Vincent Wong

Address: Department of Medicine and Therapeutics, Prince of Wales Hospital, 30-32 Ngan Shing

Street, Shatin, Hong Kong

**24-hour contact number:** +852 35054205

**Background of research** 

Non-selective beta-blockers are used in patients with cirrhosis to prevent variceal bleeding. However,

these drugs may have side effects including low blood pressure, slow heart rate, bronchospasm and

erectile dysfunction. With effective treatment of chronic liver diseases, we now know that the majority

of patients can achieve improvement or even reversal of cirrhosis. Therefore, the latest Baveno VII

consensus (published in 2022) recommends that patients with cirrhosis may stop non-selective beta-

blockers if their liver disease is well managed, the platelet count and liver stiffness measurement by

ultrasound elastography are normal, and endoscopy no longer shows the presence of varices. Although

the recommendation makes sense and may spare patients from the untoward effects of unnecessary

treatments, this practice has not been confirmed by clinical data.

Study objective

This study aims to test the feasibility and safety of stopping non-selective beta-blockers in patients

fulfilling the Baveno VII criteria.

Study procedures

Because you are an adult patient with a history of cirrhosis and are currently receiving a non-selective

beta-blocker, our centre sincerely invites you to participate in this project. You will undergo a FibroScan

examination to measure stiffness and an endoscopy to confirm the absence of varices. If both

examinations are favourable, you will stop the non-selective beta-blocker and undergo a prospective

follow-up of 5 years. At 1 year, you will undergo another endoscopy to ensure that there is no recurrence

of varices.

Baseline and follow-up visits at Months 0, 3, 6 and 12

After you have read, understood and signed this informed consent form, we will do the following:

Record your medical history and symptoms

Record your smoking habit and alcohol consumption, if any

1

- Physical examination by a doctor
- Measurement of blood pressure, pulse rate, body weight, body height, waist circumference, hip circumference, blood pressure and pulse
- Take around 10 mL of blood for blood counts, clotting, kidney and liver function
- Blood tests for hepatitis B and C virus infection (at baseline only)
- Upon your additional consent, an additional 20 mL of blood will be stored for future genetic and biochemical research
- Transient elastography to measure your liver and spleen stiffness

## **Endoscopy**

An upper gastrointestinal endoscopy will be performed at baseline and Month 12. During the procedure, you will swallow a narrow tube. The doctor will examine your oesophagus, stomach and duodenum. The doctor may also take biopsies from areas with abnormalities. The whole procedure will take around 5 to 10 minutes and does not require hospitalization.

## Long-term follow-up

After Month 12, you will resume regular follow-up at the original clinic. We will review your clinical outcomes in the next 5 years through your case records.

### **Potential risks**

Blood taking may cause pain, bruises or swelling. It may rarely cause infection or syncope. Transient elastography is a non-invasive test and will not cause any discomfort or risk. Endoscopy is a safe procedure with a less than 1% risk of bleeding, perforation and cardiorespiratory complications.

#### Other choices

Your participation is entirely voluntary. You may choose not to participate in this project. In that case, the doctor will continue you with non-selective beta-blockers.

# Charge

There is no extra charge for this study. There will not be renumeration either.

## **Confidentiality**

Your information will be kept confidential to study personnel only. As an authorised organisation, the Joint Chinese University of Hong Kong-New Territories East Cluster Clinical Research Ethics Committee may review your records to ensure that the study is conducted in an ethical manner. Your record will be stored for 15 years.

# Participant rights

You may contact Dr Vincent Wong, Principal Investigator, at +852 35054205 regarding issues of this study. You may also contact the Joint Chinese University of Hong Kong-New Territories East Cluster Clinical Research Ethics Committee at +852 35053935 regarding issues surrounding patient rights. You have the rights to refuse or stop participating in this study. Your decision will not negatively affect your future clinical care.

......

### **Informed consent**

I am aged 18 years or above and agree to participate in the above research project. I have read the Patient Information Sheet and understand the details of this project. The doctor has answered my questions satisfactorily. My participation is voluntary, and I have received a copy of the informed consent form.

I understand the benefits and risks of participating in this project. My personal information will be kept confidential. I also understand that the project was approved by the Joint Chinese University of Hong Kong-New Territories East Cluster Clinical Research Ethics Committee.

I signed this informed consent form voluntarily. I understand that I can quit this project at any time without worrying about negative consequences on my clinical care.

In addition, I agree to store my blood samples at baseline, Month 3, Month 6 and Month 12 for future genetic and biochemical studies. I understand that my decision will not affect whether I can join this study. My blood samples will be stored for 15 years.

| ☐ Agree | ☐ Do not agree |
|---------|----------------|
|---------|----------------|

| Signature | Date |
|-----------|-----------|
| Signature | Date |
| Signature | Date |
| | Signature |